CLINICAL TRIAL: NCT04421105
Title: A Phase 1,Single-centre, Randomised, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Very Low Dose LSD (5 µg, 10 µg, 20 µg) in Healthy Volunteers Aged 55-75 Years
Brief Title: A Double-blind, Placebo-controlled Study to Evaluate Very Low Dose LSD in Healthy Volunteers Aged 55-75 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eleusis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CAS-50-37-3-01
Record Dates: First submitted 2020-05-07; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 N=12 (Experimental): 6 doses at 4-day intervals for 21 days (on Study Days 1, 5, 9, 13, 17, and 21). A follow-up visit was conducted approximately 4 weeks after the last dose.
  Interventions: Drug: Lysergic acid diethylamide (LSD) 5µg
- Group 2 N=12 (Experimental): 6 doses at 4-day intervals for 21 days (on Study Days 1, 5, 9, 13, 17, and 21). A follow-up visit was conducted approximately 4 weeks after the last dose.
  Interventions: Drug: Lysergic acid diethylamide (LSD) 10µg
- Group 3 N=12 (Experimental): 6 doses at 4-day intervals for 21 days (on Study Days 1, 5, 9, 13, 17, and 21). A follow-up visit was conducted approximately 4 weeks after the last dose.
  Interventions: Drug: Lysergic acid diethylamide (LSD)20 µg
- Group 4 N=12 (Placebo Comparator): 6 doses 4-day intervals for 21 days (on Study Days 1, 5, 9, 13, 17, and 21). A follow-up visit was conducted approximately 4 weeks after the last dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lysergic acid diethylamide (LSD) 5µg
  Arms: Group 1 N=12
Drug: Lysergic acid diethylamide (LSD) 10µg
  Arms: Group 2 N=12
Drug: Lysergic acid diethylamide (LSD)20 µg
  Arms: Group 3 N=12
Drug: Placebo
  Arms: Group 4 N=12

SUMMARY:
This study was a Phase 1, double-blind, placebo-controlled, randomised study of very low dose LSD. Healthy volunteers aged 55 to 75 years with no use of LSD in the past 5 years were screened within 28 days of randomization. Subjects who met all inclusion and no exclusion criteria and provided written informed consent were randomised a 1:1:1:1 ratio to receive 6 doses of 5 µg, 10 µg, or 20 µg LSD or placebo, at 4-day intervals for 21 days (on Study Days 1, 5, 9, 13, 17, and 21). A follow-up visit was conducted approximately 4 weeks after the last dose of LSD. A total of 48 subjects were enrolled.

DETAILED DESCRIPTION:
The magnitude of the effect of LSD was explored across specific PD measures.

These included:

* Cognition and affect, including evaluation of memory, temporal perception, executive function, and learning
* Subjective effects
* Proprioception and balance

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy male or female subjects aged 55 to 75 years, inclusive (site staff endeavoured to achieve a median age of 65 years across all subjects).

  2. Subject has not been previously exposed to LSD within the past 5 years. 3. Subject is able and willing to give written informed consent, adhere to the compliance terms during participation in the study, undergo the examinations and testing set forth in the study protocol, and clearly and reliably communicate their subjective symptoms to the Investigator.

  4. A female subject is eligible to participate if she is postmenopausal (has experienced 12 consecutive months without menstruation).

  5. A male subject with a female partner is eligible to participate if he agrees to use a double barrier method of contraception. This criterion must be followed from the time of the first dose of study medication until 3 months post-last dose. Male subjects must not donate sperm for 3 months following the last dose of study medication.

Exclusion Criteria:

* General Health

  1. Subject has a history or evidence of clinically relevant psychiatric, respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders, as judged by the investigator.
  2. Subject has resting BP exceeding 160 mmHg (systolic) and 90 mmHg (diastolic), averaged across 4 assessments taken on the same day. BP measurements were taken at least 1 min apart
  3. Subject has a presence or relevant history of organic brain disorders (e.g. intracranial hypertension, impaired consciousness, lethargy, and brain tumour).
  4. Subject has a relevant history of atopy, hypersensitivity, skin allergies or allergic reactions to drugs.
  5. Subject has a clinical laboratory test result outside the reference ranges of the testing laboratory and considered clinically significant by the investigator.
  6. Subject is positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or human immunodeficiency virus I and II at screening.
  7. Subject is a current smoker. (Has not smoked for at least 1 month prior to the screening visit).
  8. Subject has a history of drug abuse/dependence in the last 12 months or has a current drug abuse/dependence, and/or is positive for drugs of abuse and alcohol tests at screening and/or baseline.
  9. Subject has a medical history that would affect the subject's safety or the study endpoints.
  10. Subject has used prescription drugs or therapy within 7 days of first dosing, unless agreed as non clinically relevant by the investigator and the Medical Monitor.
  11. Subject has used over the counter (OTC) medication or therapy, including mega-dose vitamin therapy (but excluding routine vitamins) within 7 days of first dosing, unless agreed as non clinically relevant by the investigator and the Medical Monitor.
  12. Subject has donated or received any blood or blood products within the previous 3 months prior to first dosing.
  13. Subject cannot use a computer at the required minimum level.
  14. Subject has used any investigational drug or participated in any clinical trial within 3 months of their first dosing.
  15. Subject has a current sleep disorder.
  16. Subject has a history of cataracts, active glaucoma or any other ophthalmic condition that could interfere with the eye blink assessment.
  17. Subject has a hearing loss of more than 40 dB. Subjects with > 40dB hearing loss at less than 1500Hz were excluded Subjects with > 40dB hearing loss at 1500Hz or higher can be included in the study. The hearing result from the ear with the best hearing. Provided one ear can hear at the above levels then the patient can be included.
  18. Subject has veins unsuitable for venipuncture and/or cannulation.
  19. Subject has a corrected QT interval using Fridericia's correction >450 milliseconds at any single reading.
  20. Subject is unlikely to co-operate with the requirements of the study, in the opinion of the Principal Investigator (PI) or designee.

B. Psychiatric health

1. Based on the modified SCID-CT, a subject with the lifetime presence of any of the following is excluded: psychotic symptoms that are not substance-induced or due to a medical condition or has a first- or second-degree relative with these disorders; any manic or hypomanic episode; lifetime presence of any major depressive episode; lifetime presence of substance abuse, or dependence on any substance in the past 5 years; current diagnosis of obsessive-compulsive disorder (OCD), dysthymic disorder, panic disorder, anorexia, and bulimia.
2. Subject is receiving chronic administration of tricyclic antidepressants or lithium or acute administration of selective serotonin reuptake inhibitors (SSRIs) or haloperidol, or serotonin-norepinephrine reuptake inhibitors (SNRIs) or monoamine oxidase inhibitors.
3. Subject is taking OTC doses of 5-HT or St John's Wort or Ayahuasca (which contains monoamine oxidase inhibitors in addition to dimethyltryptamine [DMT]).

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2015-11-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of very low dose LSD | 2.5 weeks
  Assessment of Adverse Events by % frequency
To evaluate the pharmacokinetics of very low dose LSD - Variation of plasma concentration over time | 12 hours
  AUC 0-12h ( pg/mL*h): area under the plasma concentration-time curve profiles from time zero to the 12 hour sample determined using the linear trapezoidal rule.
To evaluate the pharmacokinetics of very low dose LSD - Maximum Peak concentration of drug | 12 hours
  Cmax (pg/mL): maximum drug plasma concentration
To evaluate the pharmacokinetics of very low dose LSD - Half life of drug | 12 hours
  Tmax (h): time to reach maximum plasma concentration Tlag (h): time for drug to appear in plasma

SECONDARY OUTCOMES:
To evaluate the pharmacodynamic (PD) and cumulative effect of very low dose LSD on cognition. | 2.5 weeks
  The CANTAB (Cambridge Neuropsychological Test Automated Battery ) included four test that measured cognitive function. These were Reaction Time (RTI) for reaction times, Paired Associates Learning (PAL) for visual memory and learning, Rapid Visual Information Processing (RVP) for sustained memory, Spatial Working Memory (SWM) for retention of visuospatial information.
To evaluate the pharmacodynamic (PD) and cumulative effect of very low dose LSD on Acute subjective effects. | 2.5 weeks
  Assessed by the Visual Analog Scale (VAS). Items assess acute subjective drug effects (e.g. intensity, liking) Item scores are assessed on a visual scale ranging from 1% to 100%. Higher scores indicate greater subjective effects
To evaluate the pharmacodynamic (PD) and cumulative effect of very low dose LSD on the characteristics of altered states of consciousness assessed by questionnaire | 2.5 weeks
  5-Dimensional Altered States of Consciousness Questionnaire (5D-ASC). The scale ranges from no, not more than usual (on the left) to yes, very much more than usual (on the right). Items retrospectively assess subjective drug effects. Item scores are assessed on a visual scale ranging from 1% to 100%. Higher scores indicate greater subjective effects associated with a different state of consciousness
To evaluate the pharmacodynamic (PD) and cumulative effect of very low dose LSD on Balance tracking | 2.5 weeks
  Static balance as assessed by center of pressure (COP) using a portable force plate (Balance Tracking Systems, BTrackS™)
To evaluate the pharmacodynamic (PD) and cumulative effect of very low dose LSD on Proprioception | 2.5 weeks
  The ability to sense stimuli arising within the body regarding position and motion will be measured in 15 trials during which the participant will have their arm rotated to set angles and asked to reproduce the angle while blindfolded. Performance is measured as the absolute error between the target and matching angle.

OTHER OUTCOMES:
Exploratory Objective To evaluate the pharmacokinetic (PK)/PD relationship between very low dose LSD concentration and cognitive changes. | 2.5 weeks
  The relationship between LSD plasma concentration, selected PK parameters and cumulative effects of repeated LSD administration was evaluated using correlation and/or linear regression methods to evaluate possible associations with changes in cognition or affect.

CONTACTS AND LOCATIONS:
Overall Officials: Research and Development Director, Study Director — Eleusis Therapeutics

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study publication — http://link.springer.com/article/10.1007/s00213-019-05417-7